CLINICAL TRIAL: NCT00219960
Title: The Effect of North American Ginseng on Blood Pressure in Individuals With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Risk Factor Modification Centre (Other)
Collaborators: Ontario Ministry of Agriculture, Food and Rural Affairs (Other Government); Ontario Ginseng Growers Association (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RFMC-0001-77; SR-7093
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2004-06

CONDITIONS: Hypertension
Keywords: Hypertension; Blood Pressure; Ambulatory Blood Pressure Monitoring; Complementary and Alternative Medicine; Herbal; North American Ginseng; Panax Quinquefolius
MeSH Terms: conditions — Hypertension | interventions — Asian ginseng

INTERVENTIONS:
Drug: North American Ginseng (Panax Quinquefolius)

SUMMARY:
To determine the effect of North American ginseng on blood pressure in individuals with hypertension.

DETAILED DESCRIPTION:
Ginseng lacks proper clinical scrutiny for its effect on blood pressure (BP), in spite of observational evidence linking its intake to hypertension. This should be addressed considering the potential overlap between the prevalence of ginseng use and hypertension.

We undertook a single centre, randomized, controlled, double-blinded, crossover trial to determine the effect of North American ginseng (NAG) on 24-hour BP and renal function. After a 4-week placebo run-in, we randomly assigned participants to NAG or placebo treatment for 12-weeks at a dose of 3g/day. This was followed by an 8-week washout, and a subsequent 12-week period in which the opposite treatment was consumed. At run-in, and at weeks 0 and 12 of each treatment period, participants were fitted with an ambulatory BP monitor to assess 24-hour BP and serum cystatin C was measured.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 85 years
* hypertension as defined by the use of antihypertensive drugs or a seated systolic blood pressure greater than or equal to 140 mm Hg or a diastolic BP greater than or equal to 90 mm Hg at each of 3 pre-study visits.

Exclusion Criteria:

* secondary hypertension
* diabetes
* kidney
* liver disease
* unstable angina
* ginseng use for two months prior to or during the study
* any changes in the type or dose of antihypertensive drugs one month prior to or during the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52
Dates: Start 2001-04; Study Completion 2003-10

PRIMARY OUTCOMES:
Mean 24 Hour Ambulatory Blood Pressure

SECONDARY OUTCOMES:
Mean Daytime Ambulatory Blood Pressure
Mean Nighttime Ambulatory Blood Pressure
Cystatin C

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Risk Factor Modification Centre, St. Michael's Hospital
Locations (1):
- Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada